CLINICAL TRIAL: NCT04298944
Title: AuRA Study: Association of Mood With Risk for Atherosclerosis
Brief Title: Association of Mood With Risk for Atherosclerosis
Acronym: AuRA
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00226838; P50MH115842-01 (NIH)
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Mood Disorders; Hypertension; Overweight and Obesity; Vascular Stiffness; Sleep; Elevated Blood Pressure
MeSH Terms: conditions — Mood Disorders; Hypertension; Overweight; Obesity | interventions — Actigraphy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BeHealthY Cohort: Children from BeHealthY cohort who are obese/overweight but do not have mood disorders are eligible for this study. The children will be given additional questionnaires to assess emotional/behavioral well being.
  Interventions: Diagnostic Test: Cardiovascular Assessments; Diagnostic Test: Actigraphy; Diagnostic Test: Laboratory assessments; Behavioral: Emotional/ Behavioural assessments
- CHAMPION trial Cohort: Children who are overweight/obese and have severe mental illness, and who have agreed to be contacted for future research.
  Tests will be done on all participants which includes cardiovascular assessments, actigraphy, laboratory assessments and emotional/behavioral assessments.
  Interventions: Diagnostic Test: Cardiovascular Assessments; Diagnostic Test: Actigraphy; Diagnostic Test: Laboratory assessments; Behavioral: Emotional/ Behavioural assessments
- Pediatric Medical Psychiatric (PMP) Clinic Cohort: Children from the PMP Clinic who have severe mental illness but healthy weight. Tests will be done on all participants which includes cardiovascular assessments, actigraphy, laboratory assessments and emotional/behavioral assessments.
  Interventions: Diagnostic Test: Cardiovascular Assessments; Diagnostic Test: Actigraphy; Diagnostic Test: Laboratory assessments; Behavioral: Emotional/ Behavioural assessments

INTERVENTIONS:
Diagnostic Test: Cardiovascular Assessments — Participants will undergo the following cardiovascular assessments: 24-hour blood pressure monitoring, arterial stiffness measurements, endothelial function measurements.
Diagnostic Test: Actigraphy — Participants will wear an actigraph device for 7 days to measure participant's activity and sleep
Diagnostic Test: Laboratory assessments — Participants will provide blood and urine samples for laboratory assessments.
Behavioral: Emotional/ Behavioural assessments — Emotional /Behavioral well being will be determined by questionnaires: Pediatrics Adverse Childhood Experiences Questionnaire (ACEs Q), Childrens Emotion Management Scale Questionnaire (CEMS) and Behavior Assessment System for Children (BASC)

SUMMARY:
The investigators will aim to determine the association of mood disorders (MDO) with preclinical and clinical cardiovascular (CVD) risk factors among children.

The investigators will also aim to identify traditional and non traditional predictors of CVD risk among children with MDO.

DETAILED DESCRIPTION:
This research is being done to determine if mood disorders in children have an impact on stiffness of arteries and/or cause the arteries to not work as well and if MDOs impact blood pressure over a 24 hour period of time.The investigators also want to determine if children with mood disorders have any risk factors or blood tests that can predict how stiff arteries are or how well arteries function and if these are associated with cardiovascular disease risk. The investigators also want to determine if children with mood disorders have greater adverse childhood experiences, worse emotional regulation and poorer quality of sleep. The investigators hope that information from this study could help in earlier detection of cardiovascular disease risk in children.

ELIGIBILITY:
Inclusion Criteria:

* Children Ages ≤ 22 years old
* Enrolled in the CHAMPION Trial and have agreed to be contacted for future studies or children who visit PMP clinic and have MDO and a healthy weight or participants in the Be-HealthY Cohort whose data indicate no history of MDO.

Exclusion Criteria:

* Not able to speak English
* Unable to lie supine
* Significant Arrhythmia
* If participant has used vaso-active drugs the morning of the test (tobacco, caffeine decongestants, or asthma medications).

Max Age: 22 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and young adults up to 22 years of age who belong to either of the following groups:
  1. overweight/obese and no history of mood disorders
  2. overweight/obese with a mood disorder
  3. not overweight/obese with a mood disorder
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness as assessed by Pulse wave velocity | 1 day
  This will be determined from Pulse wave velocity (m/sec) done at the study visit
Arterial stiffness as assessed by Ambulatory Arterial Stiffness Index (AASI) | 1 day
  The Ambulatory Arterial Stiffness Index will be determined from data obtained from vascular measures and during 24-hour ambulatory blood pressure monitoring. Arterial stiffness increases as the regression slope approaches 0 and the AASI approaches 1.
Arterial stiffness as assessed by Augmentation Index | 1 day
  The Augmentation Index (measured as a percentage) will be determined from a vascular assessment and data obtained during 24-hour ambulatory blood pressure monitoring. A greater Augmentation Index represents a stiffer, less compliant vessel.
Endothelial function as assessed by Laser Doppler flow perfusion | 1 day
  The percent change in mean blood flow will be determined from Laser Doppler flow perfusion measurements obtained using a heating protocol.
Mean Blood pressure (mmHg) | 1 day
  Mean daytime systolic blood pressure in millimeters of mercury (mmHg) will be determined from 24-hour blood pressure monitoring.

SECONDARY OUTCOMES:
Pediatric Adverse Childhood Events (ACEs) score | 1 day
  The Pediatric ACEs questionnaire contains 17 yes or no questions about stressful or traumatic life events. Greater exposure to adverse childhood experiences (ACEs) is associated with poorer physical and mental health. Some researchers have suggested that an ACEs score of greater than or equal to 3 or 4 significantly increases the risk for health problems, however, there is no widely accepted threshold for how many ACEs endorsed is clinically significant or more predictive of these problems.
Children's Emotion Management Scale (CEMS) score | 1 day
  The Children's Emotional management scale is a questionnaire that consists of 33 questions (3 point Likert scale) examining youth's ability to regulate appropriately the youth's negative emotions (i.e. anger, sadness, and worry). Generally, poorer emotion regulation capabilities are associated with poorer health outcomes, with most research looking at CV outcomes in adults.
Behavior Assessment for Children (BASC) score | 1 day
  The Behavior Assessment for Children is a questionnaire that consists of 189 questions (True/False and 4 point Likert scale). It is a broad behavioral screening measure commonly used in child and adolescent psychology and psychiatric settings.It has three primary scales: internalizing (e.g., depression, anxiety), externalizing (e.g., aggression, hyperactivity), and total problems (combination of internalizing and externalizing plus attention problems and withdrawal subscales). Scores between 60-69 are considered "at risk" for clinical problems and scores of 70+ are considered clinically significant presence of those symptoms. Any scores that are not in this range are considered to be within normal limits and not indicative of difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy M Brady, M.D, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine Division of Pediatric Nephrology, Baltimore, Maryland, United States